CLINICAL TRIAL: NCT03701165
Title: The Effect of the DryMouth Shield on Snoring
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: VMS Medical went out of busainess
Sponsor: VMS Medical Products, Inc (Industry)
Responsible Party: Principal Investigator, Thomas Stern, MD, Medical Director, VMS Medical Products, Inc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Intervention Model Description: Cohort non-randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Snoring cohort. (Other): Subjects will undergo two nights of polysomnography. The first night will be a baseline recording. The next night subjects will use the DryMouth Shield during the polysomnography.
  Interventions: Device: DryMouth Shield

INTERVENTIONS:
Device: DryMouth Shield — The DryMouth Shield provides an elastomeric, one-piece design with breath-actuated, one-way valves configured to create an air-tight seal between the teeth and lips, which effectively reduces oral venting and air leakage while also allowing air flow into the mouth by generating a high-volume, low resistance airflow during inhalation while sealing when the user exhales.
  Other Names: Oral appliance

SUMMARY:
To measure the effect of the DryMouth Shield on snoring.

DETAILED DESCRIPTION:
The primary outcome of this study is to aid in the final design of the DryMouth Shield and to assess the effect of the DryMouth Shield on snoring frequency. To accomplish this we will compare the frequency of snores during 1) overnight polysomnography without using the DryMouth Shield and 2) overnight polysomnography using the DryMouth Shield. Secondary outcomes of the study will include: 1) compare the difference in the volume of snores without and with the use of the DryMouth Shield; 2) estimate the changes in apnea hypopnea index without and with the use of the DryMouth Shield; 3) describe symptoms of dry mouth without and with the use of the DryMouth Shield 4) describe symptoms of bruxism without and with the use of the dry mouth shield and 5) gather patient feedback about the user experience with the dry mouth shield.

ELIGIBILITY:
Inclusion Criteria:

1. reports of snoring that disturbed a bed partner or housemate and
2. an objective measure of snoring such as a previous home sleep study, lab based polysomnography, or smart phone application with a snoring index of at least 20%

Exclusion Criteria:

1. Patient's with a body mass index of greater than 35 kilogram/meter squared.
2. A history of chronic lung disease with permanently impaired lung function testing.
3. A history of cardiovascular disease including but not limited to coronary artery disease or cerebrovascular disease.
4. Current smokers.
5. Patient's with a comorbid sleep disorder including but not limited to severe sleep apnea with an apnea hypopnea index of 30 events per hour, nocturnal hypoxia necessitating oxygen, current positive airway pressure use or restless legs syndrome
6. Poor nasal patency in the judgment of the investigator
7. Use of narcotics, benzodiazepines or other respiratory suppressing medication
8. Females who are pregnant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Frequency of snoring | One night
  The percentage of number of snores during the sleep period relative to the total number of breaths during the same sleep period. A snore is defined as a breath during sleep accompanied by a vibratory noise louder than 40db

SECONDARY OUTCOMES:
Volume of snoring | One night
  The mean volume of snoring as measured by a decibel meter.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Stern, MD, Huntersville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No